CLINICAL TRIAL: NCT02595437
Title: Pharmacokinetics of Triferic (Ferric Pyrophosphate Citrate) Administered Via Dialysate and IV to Pediatric Patients on Chronic Hemodialysis
Brief Title: Triferic Pediatric Pharmacokinetic Protocol
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rockwell Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMFPC-11
Record Dates: First submitted 2015-10-30; First posted 2015-11-03 (Estimated); Results first posted 2018-10-25 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-09

CONDITIONS: End Stage Renal Disease
Keywords: dialysis; pediatric; chronic kidney disease
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic | interventions — ferric pyrophosphate; spleen fibrinolytic proteinase (human)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triferic via IV and Hemodialysate (Experimental): On study Day 1, patients will receive IV Triferic iron 0.07 mg/kg diluted in an appropriate amount of D5W administered as a 100 mL infusion into the venous return port of the blood lines during the time the patient is receiving dialysis.The rate of administration will be calculated as such that the entire amount will be administered over the course of the dialysis treatment. On study Day 3, Triferic will be mixed with the liquid bicarbonate concentrate used in the preparation of the hemodialysate solution. This will result in a final Triferic iron concentration in the dialysate of 2 µM (110 µg/L). The patients will receive Triferic via the hemodialysate over the course of the dialysis treatment.
  Interventions: Drug: Triferic

INTERVENTIONS:
Drug: Triferic
  Other Names: ferric pyrophosphate citrate; FPC

SUMMARY:
The main purpose is to determine the pharmacokinetics (PK) of Triferic iron administered intravenously in pediatric patients with chronic kidney disease on chronic hemodialysis (CKD-5HD). It is an open-label, two-period sequential dosing study.

DETAILED DESCRIPTION:
This is a Phase 1/2, open-label, 2-period, single-dose study assessing the safety and pharmacokinetics (PK) of Triferic (ferric pyrophosphate citrate, or FPC) administered via dialysate and IV to pediatric patients (< 18 years of age) receiving chronic hemodialysis (CKD-5HD).

Total participation in the study is approximately three weeks and is comprised of a screening visit, two dosing (PK) visits, and a follow-up visit.

Each patient will receive a single dose of Triferic administered IV into the venous blood return line over the duration of the dialysis. At the next scheduled dialysis session each patient will receive a single dose of Triferic administered via dialysate during a single hemodialysis session.

Blood samples will be obtained at various times to analyze for serum iron parameters and for safety.

ELIGIBILITY:
Inclusion Criteria:

A patient will be eligible for inclusion in the study only if all of the following criteria are met:

1. Parents/legal guardians of the patient have the ability to understand the requirements of the study and have demonstrated a willingness to have their child comply with all study procedures by signing an institutional review board-approved informed consent form. Where applicable, assent of the patient has also been obtained for all study procedures prior to any study-related activities.
2. Patient is <18 years of age at screening.
3. Patient has chronic kidney disease receiving in-center hemodialysis at least twice weekly for at least 1 month prior to screening.
4. Patient is receiving adequate hemodialysis as assessed by the investigator and based on a single pool Kt/V measurement >1.2.
5. Patient has a vascular access (tunneled catheter, AV fistula or AV graft) suitable to support blood flows for hemodialysis treatment.
6. Patient has a body mass of 11 lbs (5 kg).
7. Patient is iron-replete as measured by a TSAT 20% and a ferritin >100 micrograms/L at screening.
8. Patient has a whole blood Hgb concentration of 10.0 g/dL at screening.
9. If patient is receiving ESA, the dose has been stable (unchanged) for at least 3 weeks prior to Baseline admission.
10. Patient has appropriate laboratory values for their disease state at screening (per investigator judgment).
11. Patient has no significant abnormal findings on physical examination that would preclude participation in the study.
12. If the patient is female, she must be pre-pubertal, have had documented surgical sterilization prior to Baseline admission, or be practicing adequate birth control. All female patients 9 years of age and older, and also any who have reached menarche before age 9 years, must have a negative serum pregnancy test during screening. It is the investigator's responsibility to determine whether the patient has adequate birth control for study participation.

Exclusion Criteria:

A patient will not be eligible for inclusion in the study if any of the following criteria apply:

1. Patient is positive for human immunodeficiency virus (HIV) or hepatitis B by history.
2. Patient has an acute illness within 1 week of Baseline admission (patient may be screened again 2 weeks post resolution of the acute illness).
3. Patient is receiving intravenous or oral antibiotics or antifungals for any infectious process. Prophylactic antibiotics administered on a regular basis are allowed.
4. Patient has evidence of an ongoing active inflammatory process (e.g., systemic lupus erythematosus, acute or chronic active hepatitis, etc.).
5. Patient has participated in an investigational drug study within the 30 days prior to Baseline admission.
6. Administration of IV or oral iron supplements within 2 weeks prior to Baseline admission.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2015-11-01; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond D Pratt, MD FACP, Study Director — Rockwell Medical, Inc
Locations (9):
- United States (9):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Loma Linda University Hospital, Loma Linda, California
  - Lucile Packard Childrens Hospital, Stanford, California
  - Nemours/A. I. DuPont Hospital for Children, Wilmington, Delaware
  - Joe DiMagggio Children's Hospital/Memorial Regional Hospital, Hollywood, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - Childrens Mercy Hospital, Kansas City, Missouri
  - Cincinnati Children's Hospital and Medical Center, Cincinnati, Ohio
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Triferic Via IV and Hemodialysate: Triferic was administered via IV infusion on study Day 1, and then mixed with the liquid bicarbonate and administered via hemodialysate on study Day 3.
Period: Triferic Via IV
Arm/Group | Triferic Via IV and Hemodialysate
Started | 22
Completed | 21
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Triferic Via Hemodialysate
Arm/Group | Triferic Via IV and Hemodialysate
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Safety Population: All patients enrolled in the study who received any amount of Triferic, regardless of whether the dose was administered intravenously or via dialysate.
Arm/Group | Safety Population
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.8 (4.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 8
  More than one race | 0
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK) of Triferic Iron Administered IV in Pediatric CKD-5HD Patients: Cmax.
Description: The PK will be done by assessing the mean absolute and baseline-corrected Cmax of total iron with an IV infusion of Triferic at 0.07 mg iron/kg during a single dialysis session. The absolute Cmax includes the concentration of iron that was present in the serum prior to dosing as well the iron administered, while the baseline-corrected Cmax factors out the iron present in the serum prior to dosing and includes the administered iron only.
Time Frame: 0, 1, 2, 4, 4.5, 5, 6, 8, 10 hrs
Population: Pharmacokinetic Group: all patients who received at least one dose of study drug and have sufficient PK samples (a sample at the end of infusion and at least 3 samples during the elimination phase)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/deciliter
Groups:
- Triferic 0.07 mg/kg Iron Intravenous: Absolute Value: Patients were administered Triferic intravenously 0.07 mg/kg at the same time that they received their standard of care hemodialysis. The results for this group are the absolute values.
- Triferic 0.07 mg/kg Iron Intravenous: Baseline Corrected: Patients were administered Triferic intravenously 0.07 mg/kg at the same time that they received their standard of care hemodialysis. The results for this group are baseline-corrected.
Arm/Group | Triferic 0.07 mg/kg Iron Intravenous: Absolute Value | Triferic 0.07 mg/kg Iron Intravenous: Baseline Corrected
Number analyzed (Participants) | 21 | 21
microgram/deciliter | 217 (28.0) | 114 (53.7)

2. Primary Outcome: Pharmacokinetics (PK) of Triferic Iron Administered IV in Pediatric CKD-5HD Patients: AUC(Last).
Description: The PK will be done by assessing the mean absolute and baseline-corrected AUC(last) of total iron with an IV infusion of Triferic at 0.07 mg iron/kg during a single dialysis session. The absolute AUC(last) includes iron that was present in the serum prior to dosing as well the iron administered, while the baseline-corrected AUC(last) factors out the iron present in the serum prior to dosing and includes the administered iron only.
Time Frame: 0, 1, 2, 4, 4.5, 5, 6, 8, 10 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours* micrograms/ deciliters
Arm/Group | Triferic 0.07 mg/kg Iron Intravenous: Absolute Value | Triferic 0.07 mg/kg Iron Intravenous: Baseline Corrected
Number analyzed (Participants) | 21 | 21
hours* micrograms/ deciliters | 1324 (36.5) | 419 (101.6)

3. Primary Outcome: Pharmacokinetics (PK) of Triferic Iron Administered IV in Pediatric CKD-5HD Patients: AUC(0-end).
Description: The PK will be done by assessing the mean absolute and baseline-corrected AUC(0-end) of total iron with an IV infusion of Triferic at 0.07 mg iron/kg during a single dialysis session. The absolute AUC (0-end) includes iron that was present in the serum prior to dosing as well the iron administered, while the baseline-corrected AUC (0-end) factors out the iron present in the serum prior to dosing and includes the administered iron only.
Time Frame: 0, 1, 2, 4, 4.5, 5, 6, 8, 10 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours* micrograms/ deciliters
Arm/Group | Triferic 0.07 mg/kg Iron Intravenous: Absolute Value | Triferic 0.07 mg/kg Iron Intravenous: Baseline Corrected
Number analyzed (Participants) | 21 | 21
hours* micrograms/ deciliters | 648 (29.3) | 237 (76.8)

4. Secondary Outcome: Pharmacokinetics (PK) of Triferic Iron Administered Via the Hemodialysate in Pediatric CKD-5HD Patients: Cmax.
Description: The PK will be done by assessing the mean absolute and baseline-corrected Cmax of total iron. The absolute Cmax includes the concentration of iron that was present in the serum prior to dosing as well the iron administered, while the baseline-corrected Cmax factors out the iron present in the serum prior to dosing and includes the administered iron only.
Time Frame: 0, 1, 2, 4, 4.5, 5, 6, 8, 10 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/ deciliters
Groups:
- Triferic 2 Micromolar in the Hemodialysate: Absolute Value: Patients were administered Triferic at a concentration of 2 micromolar in the hemodialysate. The results for this group are the absolute values.
- Triferic 2 Micromolar in the Hemodialysate: Baseline Corrected: Patients were administered Triferic at a concentration of 2 micromolar in the hemodialysate. The results for this group are baseline-corrected.
Arm/Group | Triferic 2 Micromolar in the Hemodialysate: Absolute Value | Triferic 2 Micromolar in the Hemodialysate: Baseline Corrected
Number analyzed (Participants) | 21 | 21
micrograms/ deciliters | 261 (26.4) | 166 (54.3)

5. Secondary Outcome: Pharmacokinetics (PK) of Triferic Iron Administered Via the Hemodialysate in Pediatric CKD-5HD Patients: AUC(Last).
Description: The PK will be done by assessing the mean absolute and baseline-corrected AUC(last) of total iron. The absolute AUC (last) includes the iron that was present in the serum prior to dosing as well the iron administered, while the baseline-corrected Cmax factors out the iron present in the serum prior to dosing and includes the administered iron only.
Time Frame: 0, 1, 2, 4, 4.5, 5, 6, 8, 10 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours* micrograms/ deciliters
Groups:
- Triferic 2 Micromolar Via Hemodialysate: Absolute Value: Patients were administered Triferic at a concentration of 2 micromolar in the hemodialysate. The results for this group are the absolute values.
- Triferic 2 Micromolar Via Hemodialysate: Baseline Corrected: Patients were administered Triferic at a concentration of 2 micromolar in the hemodialysate. The results for this group are baseline-corrected.
Arm/Group | Triferic 2 Micromolar Via Hemodialysate: Absolute Value | Triferic 2 Micromolar Via Hemodialysate: Baseline Corrected
Number analyzed (Participants) | 21 | 21
hours* micrograms/ deciliters | 1453 (59.6) | 682 (82.9)

6. Secondary Outcome: Pharmacokinetics (PK) of Triferic Iron Administered Via the Hemodialysate in Pediatric CKD-5HD Patients: AUC(0-end).
Description: The PK will be done by assessing the mean absolute and baseline-corrected AUC(0-end) of total iron. The absolute AUC (0-end) includes the of iron that was present in the serum prior to dosing as well the iron administered, while the baseline-corrected Cmax factors out the iron present in the serum prior to dosing and includes the administered iron only.
Time Frame: 0, 1, 2, 4, 4.5, 5, 6, 8, 10 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours* micrograms/ deciliters
Arm/Group | Triferic 2 Micromolar Via Hemodialysate: Absolute Value | Triferic 2 Micromolar Via Hemodialysate: Baseline Corrected
Number analyzed (Participants) | 21 | 21
hours* micrograms/ deciliters | 763 (38.5) | 387 (79.6)

7. Other Pre Specified Outcome: Treatment-emergent Adverse Events (TEAEs)
Description: The incidence of treatment-emergent AEs (TEAEs) and treatment-emergent serious AEs (TESAEs) will be grouped by body system. Adverse events were recorded from study Day 1 through the following up visit (approximately 1.5 weeks).
Time Frame: 1.5 weeks
Population: Safety Population: all patients who received any amount of study medication are included in the safety population.
Measure: Count of Participants; unit: Participants
Groups:
- IV Exposure: Patients in this population had been exposed to Triferic via IV infusion only at the time of onset of the adverse event.
- IV and Hemodialysate Exposure: Patients in this population had been exposed to Triferic via the IV infusion and via hemodialysate at the time of the onset of the adverse event.
Arm/Group | IV Exposure | IV and Hemodialysate Exposure
Number analyzed (Participants) | 22 | 21
Participants | 4 | 3

ADVERSE EVENTS:
Time Frame: 1.5 weeks
Description: Adverse events were collected from date of enrollment through the date of final study visit. The total time period of collection was approximately one and a half weeks.
Groups:
- IV Exposure: Patients in this population had received Triferic via IV infusion only at the time of onset of the adverse event.
- IV and Hemodialysate Exposure: Patients in this population had received Triferic via IV infusion and via hemodialysate at the time of onset of the adverse event.
Arm/Group | IV Exposure | IV and Hemodialysate Exposure
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21
Other Adverse Events (participants affected / at risk) | 4/22 | 3/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Exposure (N=22) | IV and Hemodialysate Exposure (N=21)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Axillary Pain (General disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days